CLINICAL TRIAL: NCT01087554
Title: A Phase I Trial of Sirolimus or Everolimus or Temsirolimus (mTOR Inhibitor) and Vorinostat (Histone Deacetylase Inhibitor) in Patients With Advanced Cancer
Brief Title: Sirolimus or Everolimus or Temsirolimus and Vorinostat in Advanced Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0729; NCI-2011-00562 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-03-15; First posted 2010-03-16 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Advanced Cancer
Keywords: Advanced Cancer; Sirolimus; Rapamune; mTOR Inhibitor; Histone Deacetylase Inhibitor; Vorinostat; SAHA; Suberoylanilide Hydroxamic Acid; MSK-390; Zolinza; Everolimus; Afinitor; Zortress; RAD001; Temsirolimus; CCI-779; Torisel
MeSH Terms: interventions — Sirolimus; Vorinostat; Everolimus; temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Vorinostat + Sirolimus (Experimental): Escalation Phase: Vorinostat starting dose 100 mg by mouth on Days 7 - 28 of Cycle 1; For all other cycles, dose of 100 mg Days 1-28.
  Expansion Phase starting dose: MTD from Escalation Phase.
  Escalation Phase: Sirolimus starting dose1 mg by mouth on Days 1 - 28.
  Expansion Phase starting dose: MTD from Escalation Phase.
  Interventions: Drug: Sirolimus; Drug: Vorinostat
- Arm B: Vorinostat + Everolimus (Experimental): Escalation and Expansion Phase: Vorinostat dose 300 mg by mouth on Days 7 - 28. Rest of cycles: 300 mg by mouth on Days 1 - 28.
  Escalation Phase: Everolimus starting dose 5 mg by mouth on Days 1 - 28.
  Expansion Phase: MTD from Escalation Phase.
  Interventions: Drug: Vorinostat; Drug: Everolimus
- Arm C: Vorinostat + Temsirolimus (Experimental): Escalation and Expansion Phase: Vorinostat dose 300 mg by mouth on Days 7 - 28. Rest of cycles: 300 mg by mouth on Days 1 - 28.
  Escalation Phase: Temsirolimus starting dose 12.5 mg by vein on Days 1, 8, 15, 22.
  Expansion Phase: MTD from Escalation Phase.
  Interventions: Drug: Vorinostat; Drug: Temsirolimus

INTERVENTIONS:
Drug: Sirolimus — Escalation Phase: Sirolimus starting dose1 mg by mouth on Days 1 - 28.
  Expansion Phase starting dose: MTD from Escalation Phase.
  Other Names: Rapamune
  Arms: Arm A: Vorinostat + Sirolimus
Drug: Vorinostat — Arm A - Escalation Phase: Vorinostat starting dose 100 mg by mouth on Days 7 - 28 of Cycle 1; For all other cycles, dose of 100 mg Days 1-28.
  Expansion Phase starting dose: MTD from Escalation Phase.
  Arm B + Arm C - Escalation and Expansion Phase: Vorinostat dose 300 mg by mouth on Days 7 - 28. Rest of cycles: 300 mg by mouth on Days 1 - 28.
  Other Names: SAHA; Suberoylanilide Hydroxamic Acid; MSK-390; Zolinza
Drug: Everolimus — Escalation Phase: Everolimus starting dose 5 mg by mouth on Days 1 - 28.
  Expansion Phase: MTD from Escalation Phase.
  Other Names: Afinitor; Zortress; RAD001
  Arms: Arm B: Vorinostat + Everolimus
Drug: Temsirolimus — Escalation Phase: Temsirolimus starting dose 12.5 mg by vein on Days 1, 8, 15, 22.
  Expansion Phase: MTD from Escalation Phase.
  Other Names: CCI-779; Torisel
  Arms: Arm C: Vorinostat + Temsirolimus

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of the combination vorinostat given in combination with either sirolimus, everolimus or temsirolimus that can be given to patients with advanced cancer. The safety of this drug combination will also be studied.

The Study Drugs:

Vorinostat is designed to prevent or slow down the growth of cancer cells by blocking proteins.

Everolimus is designed to stop cells from dividing. This may stop or slow the growth or spread of cancer cells.

Temsirolimus is designed to block a protein called mTOR (a protein that is thought to cause cancer cells to grow) inside the cancer cell. This may interfere with the growth or spread of cancer cells or possibly kill them.

Sirolimus is designed to block a protein called mTOR inside the cancer cell. This may interfere with the growth or spread of cancer cells or possibly kill the cancer cells.

This is an investigational study. Sirolimus is FDA approved and commercially available as an anti-rejection drug for kidney transplant recipients. Everolimus is FDA-approved and commercially available for the treatment of pancreatic neuroendocrine tumor, subependymal giant cell astrocytoma, and renal cell carcinoma. Temsirolimus is FDA approved and commercially available for the treatment of renal cell carcinoma. Vorinostat is FDA approved and commercially available for the treatment of cutaneous T-cell lymphoma. The combination of these drugs is investigational.

Up to 249 patients will take part in this study. All will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
Study Drug Groups:

If you are found to be eligible to take part in this study, you will be assigned to a dose level of vorinostat and either sirolimus, everolimus, or temsirolimus based on when you joined this study. Up to 9 dose levels of sirolimus and vorinostat will be tested. Up to 3 dose levels of everolimus and vorinostat will be tested. Up to 3 dose levels of temsirolimus and vorinostat will be tested. Three (3) to 9 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level of the study drug combination. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of the combination vorinostat and sirolimus, everolimus, or temsirolimus is found.

Once the highest tolerated dose of the combinations are found, up to 14 participants with the tumor type that is most likely to respond to the study drug combinations will receive the study drugs at that dose level.

Study Drug Administration:

Each study "cycle" is 28 days.

There are 3 arms in this study, Arm A, Arm B, and Arm C. You will be assigned to an arm depending on when you enroll in the study and what your doctor thinks you will benefit from. You will take vorinostat either with sirolimus (Arm A), with everolimus (Arm B), or with temsirolimus (Arm C).

Everyday, you will take sirolimus by mouth 1 time a day. You should take it at about the same time each day with food and a cup (8 ounces) of water.

If you are in Arm A, on Day 7 of Cycle 1, you will start taking vorinostat by mouth 1 time a day. You should take it at about the same time each day with food and a cup (8 ounces) of water.

If your are in Arm B, you will take everolimus by mouth at the same time every day with or without food, swallowed whole with a glass (8 ounces) of water. Do not chew, break, or crush everolimus.

If you are in Arm C, you will receive temsirolimus by vein over 30-60 minutes on Days 1, 8, 15, and 22 of each cycle. You will be given standard drugs to help decrease the risk of side effects. You may ask the study staff for information about how the drugs are given and their risks.

Study Visits:

At every study visit, you will be asked about any current health conditions you have, drugs you may be taking, and if you have had any side effects.

About Days 8 and 22 of Cycle 1:

* You will have a physical exam.
* Blood (about 2 teaspoons) will be drawn for routine tests.

If you are enrolled in Arm B and have Hodgkin lymphoma, on Days 8 and 28 of Cycle 1:

* You will have a needle tumor biopsy. This biopsy will be used for DNA testing and to check for a response to the study drugs, as described above in the "Screening Tests" section.
* Blood (about 1 tablespoon) will be drawn for biomarker testing.

About Day 15 of Cycle 1, blood (about 2 teaspoons) will be drawn for routine tests.

About Day 22 of Cycles 2 and beyond:

You will have a physical exam. Blood (about 2 teaspoons) will be drawn for routine tests.

Every 4 weeks, you will have a blood (about 1 teaspoon) drawn or urine collected for a pregnancy test if you are able to become pregnant.

Every 8 weeks, you will have an x-ray, CT scan, MRI, and/or PET/CT to check the status of the disease. If the study doctor thinks it is needed, they will be performed more often.

If you are enrolled in Arm B and have Hodgkin lymphoma, at any point that the disease appears to get worse:

* You will have a needle tumor biopsy. This biopsy will be used for DNA testing and to check for a response to the study drugs, as described above in the "Screening Tests" section.
* Blood (about 1 tablespoon) will be drawn for biomarker testing.

Length of Study:

You may continue taking the study drugs for as long as you are benefitting. You will be taken off study if you experience intolerable side effects, the study doctor thinks it is in your best interest, or the disease gets worse.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a histologically-confirmed metastatic or locally advanced cancer that has failed to respond to standard therapy, progressed despite standard therapy, or for which standard therapy that increases survival by at least three months does not exist
2. There is no limit on the number of prior treatment regimens
3. Patients must be off prior cytotoxic chemotherapy for at least three weeks. For biologic or targeted therapy, there should be five half lives or three weeks, whichever is shorter, between their last treatment and the first dose on this trial.
4. Patients may receive palliative radiation therapy before or during treatment on protocol, provided that there is measurable or evaluable disease out of the radiation field. Patients may receive palliative radiation therapy, if needed, 48 hours after last dose of investigational drug. In addition patients may be enrolled on trial seven days following palliative radiation. We will closely monitor for the appearance of radiation recall reactions. Hormonal therapy may continue in patients who have been on such treatment for three months or longer.
5. ECOG performance status 0-3
6. Patients must have adequate organ and marrow function as defined by: absolute neutrophil count >/= 1000uL, platelets >/= 50,000uL, bilirubin </=2mg/dL (exceptions may apply to benign non-malignant indirect hyperbilirubinemia such as Gilbert syndrome), ALT </= 2 x ULN or </=5x ULN if liver metastases present, creatinine </= 2mg/dL
7. As the effect of sirolimus or everolimus or temsirolimus and vorinostat in combination on the developing human fetus is not known, women of child-bearing potential and men must agree to use adequate contraception (abstinence; hormonal or barrier method of birth control) for the study and at least 3 months after completion
8. Female patients with child-bearing potential must have a negative serum or urine pregnancy test within 7 days of study enrollment. Nursing mothers should discontinue nursing
9. Ability to understand and the willingness to sign a written informed consent document
10. Measurable or evaluable disease
11. Patient must be able to swallow pills

Exclusion Criteria:

1. Myocardial infarction within 3 months prior to starting treatment
2. Concomitant use of phenytoin, carbamazepine, barbiturates, rifampin, phenobarbital or St. Johns wort, cyclosporine, diltiazem, ketoconazole should be discontinued if possible. The list of CYP3A4 inhibitors: http://medicine.iupui.edu/clinpharm/ddis/clinical-table/
3. Patient has a known hypersensitivity to the components of study drugs, its analogues, or drugs of similar chemical or biologic composition
4. Patient is pregnant or breastfeeding
5. Major surgical procedure within 28 days of day 1 of therapy
6. Use of any other concurrent investigational agents or anticancer agents except for hormonal therapy as outlined in inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 249 (Estimated)
Dates: Start 2010-03 (Actual); Primary Completion 2026-08-18 (Estimated); Study Completion 2026-08-18 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 28 days
  Maximum tolerated dose (MTD) defined by dose-limiting toxicities (DLTs) that 1) occur during the first four weeks of therapy, 2) are related to the study medications (attributions: possible, probable, and likely) and 3) fulfill one of the following criteria (as graded by the NCI Common Terminology Criteria for Adverse Events). MTD is defined as highest dose level in which 6 patients have been treated with less than 2 DLTs.

SECONDARY OUTCOMES:
Tumor Response | After 4, 28 day cycles
  Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
  Progressive Disease (PD): at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
  Stable Disease (SD): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.

CONTACTS AND LOCATIONS:
Overall Officials: David S Hong, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Janku F, Park H, Call SG, Madwani K, Oki Y, Subbiah V, Hong DS, Naing A, Velez-Bravo VM, Barnes TG, Hagemeister FB, Falchook GS, Karp DD, Wheler JJ, Piha-Paul SA, Garrido-Laguna I, Shpall EJ, Fayad LE, Neelapu SS, Meric-Bernstam F, Kurzrock R, Fanale MA. Safety and Efficacy of Vorinostat Plus Sirolimus or Everolimus in Patients with Relapsed Refractory Hodgkin Lymphoma. Clin Cancer Res. 2020 Nov 1;26(21):5579-5587. doi: 10.1158/1078-0432.CCR-20-1215. Epub 2020 Oct 14. PMID 33055173
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org